CLINICAL TRIAL: NCT05914259
Title: Natural History of Chronic Kidney Disease in the US Population Using Electronic Healthcare Records
Brief Title: An Observational Study to Learn More How Chronic Kidney Disease Gradually Changes Over Time in Adults Using Electronic Healthcare Records (CKD Natural History Study)
Acronym: CKD-NH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22557
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (14):
- Diagnosed cohort - CKD Stage 1: Based on diagnosis codes (International Classification of Diseases (ICD) codes) indicating Stage 1.
  Interventions: Other: No Intervention
- Diagnosed cohort - CKD Stage 2: Based on diagnosis codes (International Classification of Diseases (ICD) codes) indicating Stage 2.
  Interventions: Other: No Intervention
- Diagnosed cohort - CKD Stage 3: Based on diagnosis codes (International Classification of Diseases (ICD) codes) indicating Stage 3.
  Interventions: Other: No Intervention
- Diagnosed cohort - CKD Stage 4: Based on diagnosis codes (International Classification of Diseases (ICD) codes) indicating Stage 4.
  Interventions: Other: No Intervention
- Diagnosed cohort - CKD Stage 5: Based on diagnosis codes (International Classification of Diseases (ICD) codes) indicating Stage 5.
  Interventions: Other: No Intervention
- Diagnosed cohort - CKD Stage Unspecified: Based on diagnosis codes (International Classification of Diseases (ICD) codes) indicating Stage Unspecified.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 1: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using Logical Observation Identifiers Names and Codes (LOINC) codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 1.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 2: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 2.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 3 overall: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 3 overall.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 3a: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 3a.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 3b: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 3b.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 4: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 4.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage 5: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage 5.
  Interventions: Other: No Intervention
- Lab based cohort - CKD Stage unspecified: Two abnormal lab measures of estimated Glomerular Filtration Rate (eGFR), or Urine Albumin-Creatinine Ratio (uACR)/ Urine Protein Creatinine Ratio (uPCR) using LOINC codes based on Kidney Disease Improving Global Outcomes (KDIGO) guidelines indicating Stage unspecified.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Following the manner of observational study, no intervention will be provided in the study.

SUMMARY:
This is an observational study in which the health data of people with chronic kidney disease are studied using electronic healthcare records. In observational studies, only observations are made without participants receiving any advice or any changes to healthcare.

Chronic kidney disease (CKD) is a condition in which the kidney's ability to work properly gradually decreases over time. This causes a buildup of waste in the body and can lead to loss of kidney function over the long term. CKD is divided into different stages based on how well the kidneys are filtering the blood.

CKD is known to increase the risk of developing serious health problems such as serious heart problems, irreversible damage to kidneys requiring either dialysis or a kidney transplant (end stage kidney disease, ESKD), and early death. However, there is limited information available about how often heart problems occur in people with different stages of CKD, and how a history of heart problems might affect future risks for CKD patients.

The purpose of this study is to collect more information on how CKD changes over time for people at different CKD stages and how it affects their heart and kidneys.

The main information that researchers will collect in this study:

changes in kidney function (worsening or improvement).

Other information that researchers will collect:

patient characteristics for each stage of CKD,

the length of time for serious heart-related conditions to occur,

the length of time it takes for CKD to progress to kidney failure,

the length of time for occurrence of deaths due to any causes, and

the length of time it takes for serious heart-related conditions and kidney failure to occur.

This study will include CKD patients above 18 years of age. Researchers will review electronic healthcare records to identify CKD patients in two ways:

using disease codes for CKD and

using lab results which show abnormal kidney function.

The data will come from participants' information stored in an electronic healthcare records database called Merative Explorys database Electronic Medical Record (EMR) in the United States of America.

The research will cover the period from January 2010 up to December 2019.

Researchers will track individual patients' data and will follow them for a maximum of 5 years or until they experience certain events like changes to their CKD stage, kidney failure, serious heart-related conditions, or death.

In this study, only available data from routine care is analyzed. No visits or tests are required.

ELIGIBILITY:
Inclusion criteria

* >18 years of age
* At least 12 months of look back period
* For Diagnosed cohorts - ICD codes for CKD diagnosis
* For Lab based cohorts - Two abnormal lab measures of eGFR or uACR/uPCR using LOINC codes.

  * Patients were included if they had the same type of test (Modification of Diet in Renal Disease (MDRD) only, CKD Epidemiology Collaboration (CKD EPI) only, Unspecified only) to estimate eGFR throughout their history because the estimation varies depending on the test used which would affect the CKD staging.

Exclusion criteria

* Birth year absent.
* Patients without any demographic information were excluded
* Patients with history of ESKD
* For Lab based cohorts:-

  * Patients were excluded if they had an incorrect test for eGFR identified by LOINC code for e.g. formula for wrong gender (Females with male MDRD formula) or wrong ethnicity (Blacks with white MDRD formula)
  * Patients with mixed types of approaches to calculate eGFR (e.g. MDRD, EPI etc.) in their history were excluded. (<20 patients)
  * We exclude lab results if the loinc code specific for ethnicity and gender does not match the patient demographics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective cohort study to assess the natural history of CKD per each CKD stage using data from Merative Explorys Electronic Medical Record (EMR) dataset in the US.
Sampling Method: Non-Probability Sample
Enrollment: 969394 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Diagnosed Cohorts - Change in CKD stage based on ICD codes | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019
Lab based Cohorts - Change in KDIFO eGFR stage based on two values and at least one of the values showing an increase or decrease by ≥25% in eGFR from baseline stage | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019

SECONDARY OUTCOMES:
Descriptive summary of patient characteristics per Chronic kidney disease (CKD) stage (1-5) | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019
Time to Major adverse coronary events (MACE)+ (composite and individual components) | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019
  MACE including all-cause mortality and also individual components (Myocardial Infarction/ Acute Coronary Syndrome (MI/ACS), Unstable Angina (UA), Coronary Artery Bypass Graft (CABG), Percutaneous Coronary Intervention (PCI), any stroke, hospitalization for heart failure)
Time to End Stage Kidney Disease (ESKD) | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019
  ESKD which includes dialysis and kidney transplant.
Time to all-cause mortality | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019
Time to MACE+ and end-stage kidney disease (ESKD) in patients who progressed or regressed | Retrospective analysis between 1 Jan 2010 to 31 Dec 2019

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Wuppertal, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.